CLINICAL TRIAL: NCT04282018
Title: A Phase 1/2, Dose Escalation and Expansion Study of BGB-10188, a Phosphatidylinositol 3-Kinase Delta (PI3Kδ) Inhibitor, Combined With Zanubrutinib in Patients With Mature B-Cell Malignancies and Combined With Tislelizumab in Patients With Solid Tumors
Brief Title: Study of BGB-10188 as Monotherapy, and in Combination With Zanubrutinib, and Tislelizumab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-3111-10188-101; CTR20220463 (Other: ChinaDrugTrials)
Record Dates: First submitted 2020-02-05; First posted 2020-02-24 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Mantle Cell Lymphoma; Diffuse Large B Cell Lymphoma; Advanced Solid Tumor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part A: BGB-10188 Monotherapy Dose Escalation (Experimental): BGB-10188 capsules administered orally once daily (QD) in 5 cohorts of escalating doses
  Interventions: Drug: BGB-10188
- Part B: BGB-10188 + Zanubrutinib Dose Escalation (Experimental): BGB-10188 capsules administered orally QD at the latest cleared dose of BGB-10188 monotherapy (Part A) in combination with zanubrutinib 160mg (2*80mg capsules) administered orally twice daily (BID)
  Interventions: Drug: BGB-10188; Drug: Zanubrutinib
- Part C: BGB-10188 + Zanubrutinib Dose Expansion (Experimental): This Part was originally planned but was cancelled by the sponsor and will not be initiated.
  Interventions: Drug: BGB-10188; Drug: Zanubrutinib
- Part D: BGB-10188 + Tislelizumab Infusion Dose Escalation (Experimental): BGB-10188 capsules administered orally QD in up to 6 cohorts of escalating doses in combination with tislelizumab 200mg IV infusion administered every 3 weeks (Q3W)
  Interventions: Drug: BGB-10188; Drug: Tislelizumab
- Part E: BGB-10188 + Tislelizumab Infusion Dose Expansion (Experimental): BGB-10188 capsules administered orally QD at two doses in combination with tislelizumab 200mg IV infusion administered Q3W
  Interventions: Drug: BGB-10188; Drug: Tislelizumab

INTERVENTIONS:
Drug: BGB-10188 — Administered as specified in the treatment arm
Drug: Zanubrutinib — Administered as specified in the treatment arm
  Other Names: BGB-3111; Brukinsa
  Arms: Part B: BGB-10188 + Zanubrutinib Dose Escalation; Part C: BGB-10188 + Zanubrutinib Dose Expansion
Drug: Tislelizumab — Administered as specified in the treatment arm
  Other Names: BGB-A317; Tevimbra; Tizveni
  Arms: Part D: BGB-10188 + Tislelizumab Infusion Dose Escalation; Part E: BGB-10188 + Tislelizumab Infusion Dose Expansion

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD), recommended dose for expansion (RDFE), safety and tolerability of BGB-10188 as monotherapy in participants with relapsed/refractory (R/R) mature B-cell malignancies; in combination with zanubrutinib in participants with R/R follicular lymphoma (FL), R/R mantle cell lymphoma (MCL) or R/R diffuse large B-cell lymphoma (DLBCL); and in combination with tislelizumab in participants with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

Parts A, B and C

1. Confirmed diagnosis of one of the following:

   * Part A: R/R CLL/SLL, R/R MZL, R/R FL, R/R MCL or R/R DLBCL
   * Part B: R/R FL, R/R MCL, or R/R DLBCL
   * Part C: R/R FL, R/R MCL, or R/R DLBCL

   CLL = chronic lymphocytic leukemia; SLL = small lymphocytic lymphoma; MZL = marginal zone lymphoma
2. Participants with MZL, FL, MCL, DLBCL, or SLL must have at least one bi-dimensionally measurable nodal lesion >1.5 cm in the longest diameter or extranodal lesion that is > 1cm in the longest diameter by computed tomography (CT) scan or magnetic resonance imaging (MRI), as defined by the Lugano Classification.

   Parts D and E
3. Part D: Histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors previously treated with standard systemic therapy (including prior chemotherapy, radiotherapy, target therapy and immunotherapy as locally, or guidance approved therapy) or for which treatment is not available or not tolerated. Enrollment will be limited to participants with advanced solid tumors for which there is clinical evidence of response to T-cell based immuno-oncology agents (eg, non-small cell lung cancer [NSCLC], small cell lung cancer [SCLC], head and neck squamous cell cancer, hepatocellular carcinoma, gastric or gastroesophageal junction carcinoma, nasopharyngeal carcinoma, renal cell carcinoma, cervical cancer, triple-negative breast cancer, ovarian cancer (OC), endometrial carcinoma, esophageal cancer, melanoma, urothelial carcinoma or participant with confirmed microsatellite instability-high [MSI-H] or mismatch repair deficient [dMMR] solid tumor, etc). Enrollment of tumor types beyond above situations requires sponsor's approval.
4. Part E: Participants with histologically or cytologically confirmed epithelial OC (including fallopian or primary peritoneal cancer) previously treated with 1 to 3 lines of systemic anticancer treatment; must be platinum resistant and checkpoint inhibitor (CPI) naïve.
5. Participants must have measurable disease as assessed by RECIST v1.1.

Key Exclusion Criteria:

Parts A, B and C

1. History of allogeneic stem-cell transplantation or chimeric antigen receptor-T (CAR-T) cell therapy.
2. For participants with DLBCL in Part A, classified as T-cell/histiocyte-rich large B-cell lymphoma, high-grade B-cell lymphoma with myelocytomatosis viral oncogene homolog and B-cell lymphoma (BCL)-2 and/or BCL-6 rearrangements, high grade B-cell lymphoma, primary mediastinal large B-cell lymphoma, Epstein-Barr virus positive DLBCL, and transformed DLBCL.

   Parts A, B, C, D and E
3. Prior exposure to PI3K inhibitor. For participants in Part B and Part C, prior exposure to BTK inhibitor and/or PI3K inhibitor.
4. Any approved anticancer therapy, including hormonal therapy, or any investigational agent or participation in another clinical study with therapeutic intent within 14 days before first dose.
5. Treatment with systemic immune-stimulatory agents (including, but not limited to, interferons and interleukin-2) within 2 weeks or 5 half-lives of the drug, whichever is later, before first dose.
6. Known human immunodeficiency virus (HIV) infection, or serologic status reflecting active viral hepatitis B (HBV) or viral hepatitis C (HCV) infection as follows:

   * HBsAg (+), or
   * HBcAb (+) and HBV DNA detected, or
   * Presence of HCV antibody. Participants with presence of HCV antibody are eligible if HCV ribonucleic acid (RNA) is undetectable

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Part A: The recommended dose for expansion (RDFE) of BGB-10188 monotherapy | Up to 8 Weeks
Part B: RDFE of BGB-10188 in combination with zanubrutinib | Up to 8 Weeks
Part D: RDFE of BGB-10188 in combination with tislelizumab | Up to 8 Weeks
Part E: Overall response rate (ORR) | Up to approximately 5 years and 6 months
  ORR is defined as the proportion of participants achieving a partial response (PR) or better
Parts A, B, D, and E: Number of participants experiencing Treatment Emergent Adverse Events (TEAEs) | Up to approximately 5 years and 6 months
Parts A, B, D, and E: Number of participants experiencing Severe Adverse Events (SAEs) | Up to approximately 5 years and 6 months
Parts A, B, D and E: Number of participants experiencing Adverse Events (AEs) Leading to Discontinuation | Up to approximately 5 years and 6 months

SECONDARY OUTCOMES:
Parts A, B, and D: Overall response rate (ORR) | Up to approximately 5 years and 6 months
  ORR is defined as the proportion of participants achieving a partial response (PR) or better
Parts B, D, and E: Duration of response (DOR) | Up to approximately 5 years and 6 months
  DOR is defined as the time from the first response documentation to the date that progression is documented after treatment initiation or death, whichever occurs first
Parts B, D, and E: Time to response (TTR) | Up to approximately 5 years and 6 months
  TTR is defined as the time from treatment initiation to the first documentation of response
Part E: Progression-free survival (PFS) | Up to approximately 5 years and 6 months
  PFS is defined as the time from treatment initiation to the first documentation of progression or death due to any cause, whichever happens first
Parts D and E: Disease control rate (DCR) | Up to approximately 5 years and 6 months
Parts A, B, D, and E: Observed maximum plasma concentration during a sample interval (Cmax) of BGB-10188 | Predose up to 7 days postdose
Parts A, B, D, and E: Area under the plasma concentration-time curve (AUC) of BGB-10188 | Predose up to 7 days postdose
Part E: Clinical Benefit Rate (CBR) | Up to approximately 5 years and 6 months
  CBR is defined as proportion of participants with best overall response, as defined by RECIST v1.1, of a CR, PR, or at least 24 weeks of stable disease
Part E: CA-125 Response Rate | Up to approximately 5 years and 6 months
  CA-125 response rate is defined as the proportion of participants achieving a CA-125 response according to the Gynecological Cancer Center Intergroup criteria; a response has occurred if there is at least a 50% reduction in CA-125 levels from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (24):
- Australia (8):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Saint Vincents Hospital Sydney, Darlinghurst, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Gallipoli Medical Research Foundation, Greenslopes, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Perth Blood Institute, West Perth, Western Australia
- China (16):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Jining No Peoples Hospital West Branch, Jining, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Zhejiang University College of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
URL: https://www.beigenemedical.com/medical-information-request